CLINICAL TRIAL: NCT03936010
Title: Replication of Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes (CANVAS Trial)
Brief Title: Replication of the CANVAS Diabetes Trial in Healthcare Claims
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-CANVAS
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Canagliflozin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- DPP4i: Reference group
  Interventions: Drug: DPP-4 inhibitor
- Canagliflozin: Exposure group
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Canagliflozin — Canagliflozin dispensing claim is exposure
  Groups: Canagliflozin
Drug: DPP-4 inhibitor — DPP4 inhibitor dispensing claim is reference
  Groups: DPP4i

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates: 4/1/2013-12/31/2016 (market availability of sitagliptin in the U.S. started on 10/17/2006). For Optum, 4/1/2013-9/30/2017.

Inclusion Criteria:

* Man or woman with a diagnosis of type 2 diabetes with glycated hemoglobin level ≥7.0% to≤10.5% at screening and be either

  1. not currently on antihyperglycemic agent (AHA) therapy or
  2. on AHA monotherapy or combination therapy with any approved class of agents: e.g., sulfonylurea, metformin, peroxisome proliferator-activated receptor gamma (PPARγ) agonist, alpha-glucosidase inhibitor, glucagon-like peptide-1 (GLP-1) analogue, dipeptidyl peptidase-4 (DPP-4) inhibitor, or insulin.
* Age ≥30 years with documented symptomatic atherosclerotic cardiovascular disease
* Age ≥50 years with 2 or more of the following risk factors determined at the screening visit

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes, pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy.
* History of one or more severe hypoglycemic episode within 6 months before screening
* Ongoing, inadequately controlled thyroid disorder.
* Renal disease that required treatment with immunosuppressive therapy or a history of dialysis or renal transplant.
* MI, unstable angina, revascularization procedure, or cerebrovascular accident within 3 months before screening, or a planned revascularization procedure, or history of New York Heart Association (NYHA) Class IV cardiac disease.
* Findings on 12-lead electrocardiogram (ECG) that would require urgent diagnostic evaluation or intervention
* History of hepatitis B surface antigen or hepatitis C antibody positive
* Any history of or planned bariatric surgery.
* History of malignancy within 5 years before screening
* History of human immunodeficiency virus (HIV) antibody positive.
* Subject has a current clinically important hematological disorder (e.g., symptomatic anemia, proliferative bone marrow disorder, thrombocytopenia).
* Major surgery (i.e., requiring general anesthesia) within 3 months of the screening visit or any surgery planned during the subject's expected participation in the study
* Current use of other sodium glucose co-transporter 2 (SGLT2) inhibitor.
* Current use of a corticosteroid medication or immunosuppressive agent, or likely to require treatment with a corticosteroid medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing canagliflozin to the DPP-4 inhibitor (DPP4i) antidiabetic class. DPP4is serve as a proxy for placebo, since this class of antidiabetic drugs is not known to have an impact on the outcome of interest. The comparison against DPP4 inhibitors is the primary comparison. Initiators of 2nd generation sulfonylureas are used as a secondary comparator group. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of canagliflozin or a comparator drug (cohort entry date). Follow-up for the outcome (3P-MACE), begins the day after drug initiation. As in the trial, patients are allowed to take other antidiabetic medications during the study.
Sampling Method: Non-Probability Sample
Enrollment: 152202 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Relative hazard of composite outcome of Stroke, MI, and Mortality | Through study completion (a median of 120-140 days)
  Relative hazard of composite outcome of MI, stroke, and mortality - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Womens
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Franklin JM, Patorno E, Desai RJ, Glynn RJ, Martin D, Quinto K, Pawar A, Bessette LG, Lee H, Garry EM, Gautam N, Schneeweiss S. Emulating Randomized Clinical Trials With Nonrandomized Real-World Evidence Studies: First Results From the RCT DUPLICATE Initiative. Circulation. 2021 Mar 9;143(10):1002-1013. doi: 10.1161/CIRCULATIONAHA.120.051718. Epub 2020 Dec 17. PMID 33327727

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT03936010/Prot_SAP_002.pdf